CLINICAL TRIAL: NCT05403541
Title: A Phase 3, Multi-center, Randomized, Quadruple-blind, Placebo-controlled Study to Assess the Efficacy and Safety of Batoclimab as Induction and Maintenance Therapy in Adult Participants With Generalized Myasthenia Gravis (gMG)
Brief Title: Phase 3 Study to Assess the Efficacy and Safety of Batoclimab as Induction and Maintenance Therapy in Adult Participants With Generalized Myasthenia Gravis
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Immunovant Sciences GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IMVT-1401-3101
Record Dates: First submitted 2022-05-26; First posted 2022-06-03 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Generalized Myasthenia Gravis
Keywords: monoclonal antibody; batoclimab; IMVT-1401; Myasthenia Gravis; acetylcholine receptor; RVT-1401
MeSH Terms: conditions — Myasthenia Gravis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Sponsor Staff is also masked, so the study is Quadruple-blind.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Batoclimab Induction Dose 1 (Period 1) (Experimental)
  Interventions: Drug: Batoclimab 680 mg SC weekly
- Batoclimab Induction Dose 2 (Period 1) (Experimental)
  Interventions: Drug: Batoclimab 340 mg SC weekly
- Placebo Induction Dose (Period 1) (Placebo Comparator)
  Interventions: Drug: Matching Placebo SC
- Batoclimab Maintenance Dose 1 (Period 2) (Experimental)
  Interventions: Drug: Batoclimab 340 mg SC weekly
- Batoclimab Maintenance Dose 2 (Period 2) (Experimental)
  Interventions: Drug: Batoclimab 340 mg SC bi-weekly
- Placebo Maintenance Dose (Period 2) (Placebo Comparator)
  Interventions: Drug: Matching Placebo SC

INTERVENTIONS:
Drug: Batoclimab 680 mg SC weekly — Batoclimab is a fully human anti-neonatal fragment crystallizable receptor (FcRn) monoclonal antibody
  Other Names: IMVT-1401
  Arms: Batoclimab Induction Dose 1 (Period 1)
Drug: Batoclimab 340 mg SC weekly — Batoclimab is a fully human anti-neonatal fragment crystallizable receptor (FcRn) monoclonal antibody
  Other Names: IMVT-1401
  Arms: Batoclimab Induction Dose 2 (Period 1); Batoclimab Maintenance Dose 1 (Period 2)
Drug: Matching Placebo SC — Placebo
  Arms: Placebo Induction Dose (Period 1); Placebo Maintenance Dose (Period 2)
Drug: Batoclimab 340 mg SC bi-weekly — Batoclimab is a fully human anti-neonatal fragment crystallizable receptor (FcRn) monoclonal antibody
  Other Names: IMVT-1401
  Arms: Batoclimab Maintenance Dose 2 (Period 2)

SUMMARY:
The purpose of this 4-period study is to confirm the efficacy and safety of batoclimab in participants with gMG. In Period 1, participants will be randomized 1:1:1 to receive batoclimab 680 milligrams (mg) subcutaneously (SC) once a week (QW) or 340 mg SC QW or placebo. The primary efficacy endpoint will be assessed by change in the myasthenia gravis activities of daily living (MG- ADL) score in acetylcholine receptor antibody seropositive (AChRAb+) participants. In Period 2, participants previously treated with batoclimab will be re-randomized to stay on batoclimab (340 mg SC QW or 340 mg SC every two weeks) or receive placebo treatment. The secondary endpoint of maintenance of efficacy will be assessed by change in the MG- ADL score in AChRAb+ participants. Participants demonstrating a response to batoclimab during either Period 1 or 2 may enter the long-term extension (Period 3). Participants who complete Period 3 are eligible to participate in Period 4 (Optional Long-Term extension) according to their treatment assignment in Period 3.

ELIGIBILITY:
Inclusion Criteria:

1. Are ≥ 18 years of age at the Screening Visit.
2. Have mild to severe gMG by Myasthenia Gravis Foundation of America (MGFA) classification Class II, III, or IVa at the Screening Visit.
3. Have a QMG score ≥ 11 at the Screening and Baseline Visits.
4. Have a MG-ADL score of ≥ 5 at the Screening and Baseline Visits.
5. Additional inclusion criteria are defined in the protocol.

Exclusion Criteria:

1. Have experienced myasthenic crisis within 3 months of the Screening Visit.
2. Have had a thymectomy performed < 6 months prior to the Screening Visit or have a planned thymectomy during the study period.
3. Have any active or untreated malignant thymoma.
4. Have received any agent or therapy (exclusive of those identified within inclusion criteria) with immunosuppressive properties (e.g., stem cell therapy, chemotherapies) within the past year.
5. Have used anti-FcRn treatment within 3 months prior to the Screening Visit or have a documented history of non-response to prior anti-FcRn treatment.
6. Additional exclusion criteria are defined in the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2022-06-27 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Myasthenia Gravis Activities of Daily Living (MG-ADL) score in acetylcholine receptor (AChR) Ab seropositive (AChRAb+) participants | Baseline (Day 1) to Week 12
  MG-ADL is an 8-item, participant-reported questionnaire that assesses gMG symptoms and their effects on activities of daily living. Each item is assessed on a 4-point scale where a score of 0 represents normal function and a score of 3 represents loss of ability to perform that function. Total score ranges from 0 to 24, with higher scores indicating greater functional impairment and disability.

SECONDARY OUTCOMES:
Change from Baseline in Quantitative Myasthenia Gravis (QMG) score in AChRAb+ participants | Baseline (Day 1) to Week 12
  QMG is clinician-reported assessment to evaluate muscle weakness in participants with MG. The QMG consists of 13 items ranging from 0 to 3 with 3 being the most severe. Total score ranges from 0 to 39, with higher scores representing greater impairment.
Change from Baseline in MG-ADL score for AChRAb+ randomized withdrawal participants | Baseline (Week 12) to Week 24
Percentage of AChRAb+ participants with greater than equal to (>=) 3-point improvement in QMG score | Up to Week 12
Percentage of AChRAb+ participants achieving MG-ADL score of 0 or 1 by Week 12 | Up to Week 12
Change from Baseline in MG-ADL score in AChRAB- (AChRAB negative) participants | Baseline (Day 1) to Week 12
Percentage of Participants with Treatment Emergent Adverse Events (TEAEs) | Up to 76 Weeks
  An adverse event (AE) is defined as any untoward medical occurrence in a participant who has either been administered a study drug or has undergone study procedures.
Percentage of Participants With Clinically Significant Changes in Vital Sign Measurements | Up to 76 Weeks
  Vital signs, including systolic and diastolic blood pressures, pulse rate, respiratory rate, and temperature will be obtained and recorded at specified timepoints. All vital sign measures will be obtained with the participant in the supine position and having rested for at least 5 minutes.
Number of Participants with Clinically Significant Changes in Laboratory Results | Up to 76 Weeks
  Blood samples will be collected at specified timepoints for the analysis of laboratory parameters including clinical chemistry, hematology and urinalysis.
Percentage of participants with clinical laboratory-related TEAEs or treatment emergent laboratory abnormalities. | Up to 76 Weeks

CONTACTS AND LOCATIONS:
Locations (105):
- United States (33):
  - Site Number -1022, Phoenix, Arizona
  - Site Number -1029, Scottsdale, Arizona
  - Site Number -1002, Carlsbad, California
  - Site Number -1009, Irvine, California
  - Site Number - 1012, Olive View, California
  - Site Number -1032, San Francisco, California
  - Site Number - 1027, Aurora, Colorado
  - Site Number - 1025, New Haven, Connecticut
  - Site Number -1017, Boca Raton, Florida
  - Site Number -1007, Clearwater, Florida
  - Site Number -1010, Maitland, Florida
  - Site Number - 1020, Miami, Florida
  - Site Number -1019, Orlando, Florida
  - Site Number - 1028, Port Charlotte, Florida
  - Site Number - 1015, Tampa, Florida
  - Site Number -1011, Fairway, Kansas
  - Site Number -1003, Lexington, Kentucky
  - Site Number -1013, East Lansing, Michigan
  - Site Number - 1024, Minneapolis, Minnesota
  - Site Number - 1021, Buffalo, New York
  - Site Number - 1018, Chapel Hill, North Carolina
  - Site Number - 1008, Durham, North Carolina
  - Site Number -1004, Cleveland, Ohio
  - Site Number -1006, Portland, Oregon
  - Site Number - 1023, Philadelphia, Pennsylvania
  - Site Number - 1030, Charleston, South Carolina
  - Site Number - 1026, Memphis, Tennessee
  - Site Number -1001, Austin, Texas
  - Site Number -1016, Dallas, Texas
  - Site Number - 1034, Houston, Texas
  - Site Number - 1014, Round Rock, Texas
  - Site Number -1031, Murray, Utah
  - Site Number -1005, Charlottesville, Virginia
- Argentina (3):
  - Site Number - 5002, Buenos Aires
  - Site Number - 5001, Buenos Aires
  - Site Number - 5003, Rosario
- Brazil (2):
  - Site Number - 5501, Ribeirão Preto
  - Site Number- 5503, Rio de Janeiro
- Canada (4):
  - Site Number -2001, Edmonton, Alberta
  - Site Number - 2003, Vancouver, British Columbia
  - Site Number - 2002, Toronto, Ontario
  - Site Number - 2004, Montreal, Quebec
- Georgia (5):
  - Site Number -8002, Tbilisi
  - Site Number -8004, Tbilisi
  - Site Number -8001, Tbilisi
  - Site Number -8003, Tbilisi
  - Site Number - 8005, Tbilisi
- Germany (6):
  - Site Number - 6507, Berlin
  - Site Number - 6506, Bochum
  - Site Number - 6501, Hamburg
  - Site Number - 6503, Jena
  - Site Number -6504, Leipzig
  - Site Number -6502, Würzburg
- Hungary (2):
  - Site Number -7553, Budapest
  - Site Number - 7552, Kistarcsa
- Italy (7):
  - Site Number - 6004, Bergamo
  - Site Number -6006, Brescia
  - Site Number - 6002, Genova
  - Site Number - 6003, Milan
  - Site Number - 6007, Napoli
  - Site Number -6001, Napoli
  - Site Number -6005, Roma
- Japan (20):
  - Site Number - 4020, Asahikawa-shi
  - Site Number - 4014, Fuchu-shi
  - Site Number - 4002, Hanamaki-shi
  - Site Number - 4013, Higashimatsushima
  - Site Number - 4006, Kagawa
  - Site Number - 4009, Kawasaki-shi
  - Site Number - 4012, Koriyama-shi
  - Site Number - 4007, Koshigaya-shi
  - Site Number - 4011, Matsuyama
  - Site Number - 4008, Miyagi
  - Site Number - 4003, Narita-shi
  - Site Number - 4010, Osaka
  - Site Number - 4004, Osaka
  - Site Number - 4001, Osaka
  - Site Number - 4005, Tokyo
  - Site Number - 4018, Toyama
  - Site Number - 4016, Yokohama
  - Site Number - 4019, Yokohama
  - Site Number - 4015, Yokohama
  - Site Number - 4017, Yonago-shi
- Site Number - 2601, Mexico City, Mexico
- Poland (8):
  - Site Number - 3007, Gdansk
  - Site Number -3001, Katowice
  - Site Number -3004, Krakow
  - Site Number - 3003, Krakow
  - Site Number -3002, Krakow
  - Site Number - 3008, Lublin
  - Site Number -3006, Poznan
  - Site Number - 3005, Warsaw
- Romania (3):
  - Site Number -7502, Constanța
  - Site Number -7501, Târgu Mureş
  - Site Number -7503, Timișoara
- Serbia (2):
  - Site Number - 9001, Belgrade
  - Site Number - 9002, Niš
- South Korea (2):
  - Site Number -4505, Daegu
  - Site Number -4501, Seoul
- Spain (5):
  - Site Number -3502, Barcelona
  - Site Number -3505, Barcelona
  - Site Number -3504, Córdoba
  - Site Number -3501, Madrid
  - Site Number -3503, Madrid
- United Kingdom (2):
  - Site Number - 7001, Liverpool
  - Site Number - 7002, Sheffield

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Benatar M, Wiendl H, Nowak R, Zheng Y, Macias W. Batoclimab as induction and maintenance therapy in patients with myasthenia gravis: rationale and study design of a phase 3 clinical trial. BMJ Neurol Open. 2024 Jan 10;6(1):e000536. doi: 10.1136/bmjno-2023-000536. eCollection 2024. PMID 38268752